CLINICAL TRIAL: NCT03485547
Title: Phase 1 Study of Venetoclax, a BCL2 Antagonist, for Patients With Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Brief Title: Study of Venetoclax, a BCL2 Antagonist, for Patients With Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Andrew Lane, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-045
Record Dates: First submitted 2018-03-27; First posted 2018-04-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm
Keywords: Blastic Plasmacytoid Dendritic Cell Neoplasm; BPDCN
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax (Experimental): * Venetoclax is administered on a daily basis orally.
  * The investigators will use a modified 3+3 with a de-escalation dose level design to establish the appropriate and tolerable dose of venetoclax.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — VENCLEXTA targets BCL-2 in order to help restore the process of apoptosis. Through apoptosis, your body allows cancer cells and normal cells to self-destruct
  Other Names: Venclexta

SUMMARY:
This research study is studying a drug as a possible treatment for BPDCN.

The intervention involved in this study is: Venetoclax

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the safest dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved venetoclax for this specific disease but it has been approved for other uses.

Based on laboratory data where it was found that BPDCN cells die after treatment with Venetoclax, the investigators believe that this drug will be effective in treating patients with BPDCN.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of blastic plasmacytoid dendritic cell neoplasm (BPDCN) per 2016 WHO criteria
* Age > 18 years
* In Stage 1 (modified 3+3): BPDCN relapsed after or refractory to at least one prior treatment regimen (hydroxyurea is not considered a prior treatment regimen)
* In Stage 2 (expansion):

  * (A) BPDCN relapsed after or refractory to at least one prior treatment regimen (hydroxyurea is not considered a prior treatment regimen)

    ---OR
  * (B) Treatment-naïve BPDCN, and age > 75 years; or treatment-naïve BPDCN, and age > 18 years and who decline intensive induction chemotherapy or who are unfit due to co-morbidity or other factors (see APPENDIX A for unfitness definitions)
* ECOG performance status 0, 1, or 2
* Adequate organ function as defined by:

  * Serum creatinine < 1.5x ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x ULN
  * Total bilirubin < 1.5x ULN (if total bilirubin is > 1.5x but < 3x ULN, and thought to be elevated due to Gilbert's disease or the patient's BPDCN, the subject may be eligible but must discuss with the PI)
* Ability to understand and the willingness to sign a written informed consent document.
* Able to adhere to study visit schedule and other protocol requirements including follow-up for survival assessment
* Women of child-bearing potential and men enrolled on this protocol must agree to use adequate contraception for the duration of study participation and for 2 months after completion venetoclax administration.

Exclusion Criteria:

* Prior treatment with venetoclax
* Received treatment with chemotherapy, radiation, or biologic cancer therapy within 14 days of first protocol treatment. Prior and concurrent hydroxyurea is permitted during the first cycle.
* Hematopoietic stem cell transplantation (HSCT) within 60 days of first protocol treatment, or receipt of immunosuppressive therapy for graft-versus-host disease treatment or prophylaxis within 14 days of first protocol treatment, or active graft-versus-host-disease
* Known active CNS involvement by BPDCN
* Known positive status for HIV infection; known active hepatitis B or hepatitis C infection
* Clinically significant cardiopulmonary disease including uncontrolled or NYHA class 3 or 4 congestive heart failure, uncontrolled angina, uncontrolled hypertension, uncontrolled arrhythmia, myocardial infarction or stroke within 6 months of first protocol treatment
* Patients with known active advanced malignant solid tumors are excluded (except for basal or squamous skin cancers, or carcinomas in situ). Patients with additional hematologic malignancies that require treatment are excluded.
* Patients with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in the developing fetus with venetoclax (negative urine or serum pregnancy test required within 14 days of Cycle 1, Day 1). Because nursing infants have unknown potential for adverse events secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with venetoclax.
* Infection is a common feature of BPDCN and acute leukemias. Patients with active infection are permitted to enroll provided that the infection is controlled (patients on IV or PO antibiotics are allowed). Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.
* Subject has received the following within 7 days prior to the initiation of study treatment:

  * Strong and moderate CYP3A inducers
  * Strong and moderate CYP3A inhibitors
* Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or Star fruit within 3 days prior to the initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 2 years

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
Complete Response | 2 years
Partial Response | 2 years
Overall Survival | 2 years
Progression free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lane, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang SY, Thomassen K, Kurch L, Opitz S, Franke GN, Bach E, Platzbecker U, Kayser S. Combination of Tagraxofusp and Azacitidine Is an Effective Option for Relapsed Blastic Plasmacytoid Dendritic Cell Neoplasm After Allogeneic Hematopoietic Stem-Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Jul;21(7):e579-e582. doi: 10.1016/j.clml.2021.02.008. Epub 2021 Mar 2. No abstract available. PMID 33795208